CLINICAL TRIAL: NCT02335619
Title: Early Integrated Supportive Care Study for Gastrointestinal Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pippa Hawley (Other)
Responsible Party: Sponsor-Investigator, Pippa Hawley, Head Palliative Care Physician, British Columbia Cancer Agency
Organization: British Columbia Cancer Agency (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H14-02082
Record Dates: First submitted 2015-01-07; First posted 2015-01-12 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Palliative Care (Active Comparator): During their first oncology appointment, the intervention arm patients will self-report any symptoms related to their cancer or treatment to the study team; scores at or above a defined benchmark will be seen by Pain and Symptom Management/Palliative Care team members during or immediately after their oncology appointment. Patients will be asked to self-report symptoms once a month following recruitment, for 4 months.
  Interventions: Behavioral: Early palliative care
- Standard Care (No Intervention): During their first oncology appointment, the control arm patients will self-report any symptoms related to their cancer or treatment to the study team; self-reports will be collected but not shared with the Pain and Symptom Management/Palliative Care team, and patients will continue with their oncology appointment as per standard procedure. Patients will be asked to self-report symptoms once a month following recruitment, for 4 months.

INTERVENTIONS:
Behavioral: Early palliative care
  Arms: Early Palliative Care

SUMMARY:
Currently at the BC Cancer Agency, oncologists decide when to refer a patient to the Pain and Symptom Management/Palliative Care (PSMPC) team, and their decisions are made subjectively and without standard guidelines/symptom assessment tools. Patients are often referred late in their treatment. The PSMPC team sees patients in their own clinic, separately from the oncologists, and do not often collaborate in a patient's care.

Early integration of palliative care into oncological care has been shown to improve quality of life and to prolong survival, as well as to reduce inappropriately aggressive oncological care at end of life, and reduce costs of care. We will test an early oncology-integrated palliative care model, with the aims of determining whether 1) the introduction of PSMPC support at the time of diagnosis leads to better symptom management and quality of life of patients, 2) early integration of palliative care into medical oncology care reduces aggressiveness of cancer treatment near end of life, and 3) a fully integrated service delivery model is sustainable.

DETAILED DESCRIPTION:
Gastrointestinal (GI) medical oncologists will be assigned to intervention or control groups, according to whether or not they have clinics scheduled on 2 specific half days each week, to coincide with PSMPC clinics. New patients attending the specified clinics under each oncologist will be automatically fall under whichever group their oncologist has been assigned. Control patients will be those seen at clinics other than the 2 specified intervention clinics.

Patients will be approached for study participation in the waiting room of the GI clinic as they await their first oncology appointment. Those who agree to participate will be asked to complete a symptom assessment questionnaire at baseline and once a month for 4 months. This timing is meant to coincide with their regularly scheduled follow up appointments with the GI oncologist.

Symptom scores from the completed assessment forms will be entered into a study database, created with the BC Cancer Agency IDs of the study participants alongside an anonymized study ID.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with a gastrointestinal (GI) cancer
* have appointments in GI clinic during study days
* able to complete a symptom assessment form on their own or with the help of a family member or interpreter

Exclusion Criteria:

* already receiving care from the Pain and Symptom Management/Palliative Care team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2015-02; Primary Completion 2018-12 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Total symptom distress score | 4 months after recruitment
  Total symptom distress score will be measured using a modified Edmonton Symptom Assessment System (ESAS). Individual patient scores at 4 months will be compared to their scores at recruitment (first oncology appointment).

SECONDARY OUTCOMES:
Use of health services | 4 months after recruitment
  This outcome will be evaluated by measuring the following within each treatment group:
  number of hospital admissions for non-treatment reasons; number of emergency room visits; number of referrals to the Pain and Symptom Management/Palliative Care team; number of Pain and Symptom Management/Palliative Care follow up visits per patient
Aggressiveness of cancer treatment | 4 months after recruitment
  This outcome will be evaluated by measuring the following within each treatment group:
  number of patients being treated with chemotherapy in last 2-4 weeks of life; number of patients admitted to home hospice in last 3-14 days of life
Details of death (survival time from first oncology appointment at BC Cancer location of death (home, hospice, Cancer Centre) | 1 year from recruitment
  This data will be collected for those patients who do not survive past one year of recruitment. The outcome will be evaluated by the following:
  survival time from first oncology appointment at BC Cancer location of death (home, hospice, Cancer Centre)

CONTACTS AND LOCATIONS:
Overall Officials: Philippa Hawley, B.Med, Principal Investigator — British Columbia Cancer Agency
Locations (1):
- British Columbia Cancer Agency - Vancouver Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT02335619/Prot_SAP_000.pdf